CLINICAL TRIAL: NCT04556526
Title: A Phase 3 Open-label Randomized Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of a 2-dose Ebola Vaccine Regimen of Ad26.ZEBOV Followed by MVA-BN-Filo in Healthy Pregnant Women
Brief Title: A Study of a 2-dose Ebola Vaccine Regimen of Ad26.ZEBOV Followed by MVA-BN-Filo in Healthy Pregnant Women
Acronym: INGABO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Center for Family Health Research (CFHR) (Unknown); Coalition for Epidemic Preparedness Innovations (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR108739; VAC52150EBL3010 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Ad26.ZEBOV, MVA-BN-Filo (Experimental): Participants will receive intramuscular (IM) injection (0.5 milliliter [mL]) of Adenovirus serotype 26 encoding the ebola virus mayinga glycoprotein (Ad26.ZEBOV) as Dose 1 (5*10^10 viral particle(s) [vp]) on Day 1, followed by modified vaccinia Ankara Bavarian Nordic vector encoding multiple filovirus proteins (MVA-BN-Filo) as Dose 2 (1*10^8 infectious unit(s) [Inf U]) on Day 57.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo
- Group B: No vaccination during pregnancy (Other): Participants (pregnant women) in control Group B will not receive any vaccination during pregnancy. However, women in this group will receive the 2-dose vaccination regimen at the earliest 6 weeks after delivery/termination of pregnancy that is Dose 1 of Ad26.ZEBOV vaccine (0.5 mL) (5*10^10 vp) on Day 1 by IM injection followed by 0.5 mL of MVA-BN-Filo (1*10^8 Inf U) vaccine by IM injection 56 days after Dose 1.
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo

INTERVENTIONS:
Biological: Ad26.ZEBOV — Participants in Group A will receive 0.5 mL IM injection of Ad26.ZEBOV vaccine. Participants in Group B will receive Ad26.ZEBOV 6 weeks after delivery/termination of pregnancy.
Biological: MVA-BN-Filo — Participants in Group A will receive 0.5 mL IM injection of MVA-BN-Filo vaccine. Participants in Group B will receive MVA-BN-Filo 6 weeks after delivery/termination of pregnancy.

SUMMARY:
The purpose of this study is: a) to assess adverse maternal/fetal outcomes in pregnant women randomized to receive the 2- dose Ebola vaccine regimen (Ad26.ZEBOV, MVA-BN-Filo [Group A]) and in control women (unvaccinated pregnant women [Group B]); and b) to assess adverse neonatal/infant outcomes in neonates/infants born to women randomized to receive the 2-dose Ebola vaccine regimen (Ad26.ZEBOV, MVA-BN-Filo [Group A]) and in neonates/infants born to control women (unvaccinated during pregnancy [Group B]).

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, obstetric history, and vital signs performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening
* Confirmed singleton pregnancy by positive urine human chorionic gonadotropin (HCG) and ultrasound at time of screening and informed consent, and reconfirmed pregnancy via ultrasound at Randomization/Day 1
* Residing within catchment area of the study site
* Evidence of normal progress of gestation prior to Randomization (Day 1) based on obstetric evaluation (including obstetric history, obstetric examination and fetal ultrasound)

Exclusion Criteria:

* History of Ebola Virus Disease (EVD) (self-declared or laboratory confirmed)
* Has received any experimental candidate Ad26- or MVA-based vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines [for example, polysorbate 80, ethylenediaminetetraacetic acid (EDTA) or L-histidine for Ad26.ZEBOV vaccine; tris (hydroxymethyl)-amino methane (THAM) for MVA-BN-Filo vaccine]), including known allergy to egg, egg products, chicken proteins and aminoglycosides
* Participant with acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or body temperature greater than or equal to (>=)38.0ºC on Day 1 will be excluded from enrollment at that time but may be rescheduled for enrollment at a later date
* During the 6 weeks prior to screening, have had any of (a) confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (COVID-19) infection (test positive), OR (b) suspected SARS-CoV-2 infection (clinical features without documented test results), OR (c) close contact with a person with known or suspected SARS-CoV-2 infection
* Obstetric history including: a. >= 2 consecutive spontaneous abortions, b. history of pre-eclampsia or eclampsia, c. rhesus negative multigravida, d. grand multigravida (greater than [>] 5 previous pregnancies, e. previous late still birth (defined as loss of pregnancy at any time after 28 weeks gestation), f. previous low birth weight baby or premature delivery (defined as a delivery before 37 weeks gestation), g. previous neonatal death (defined as death of an infant within the first 28 days of life), h. previous delivery of an infant with a known or suspected genetic or chromosomal abnormality, i. history of other significant pregnancy-related or neonatal complications judged likely to affect the safety of the mother or infant or to significantly compromise the endpoint data collected

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4031 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Maternal Deaths | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with maternal deaths will be reported. Maternal death is the death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.
Percentage of Participants with Spontaneous Abortion | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with spontaneous abortion will be reported. Spontaneous abortion is a pregnancy loss that occurs up to 21 weeks 6 days of gestation.
Percentage of Participants with Stillbirth | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with stillbirth will be reported. Stillbirth is fetal death at or after 21 weeks 6 days of gestation.
Percentage of Participants on the Pathways to Preterm Birth | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants on the pathways to preterm birth will be reported. Pathways to preterm birth is a clinical syndrome characterized by any one or some combination of the following four pathways: 1) Premature preterm rupture of membranes, 2) Preterm labor, 3) Insufficient cervix, 4) Provider- initiated preterm birth.
Percentage of Participants with Pre-eclampsia/ eclampsia | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with pre-eclampsia/ eclampsia will be reported. Pre-eclampsia is new-onset or worsening of existing hypertension with new-onset proteinuria after 20 weeks gestation.
Percentage of Participants with Antenatal Bleeding | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with antenatal bleeding will be reported. Antenatal bleeding is vaginal or suspected intrauterine, intraperitoneal, or retroperitoneal bleeding in the second or third trimester of pregnancy.
Percentage of Participants with Postpartum Hemorrhage | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with postpartum hemorrhage will be reported. Postpartum hemorrhage is genital bleeding after delivery estimated at 1000 ml or more, or leading to hypotension or blood transfusion, or leading to severe maternal outcome (maternal death or maternal near miss) as defined by World Health Organization (WHO).
Percentage of Newborns with Major Congenital Malformations born to Participants | At birth
  Percentage of newborns with major congenital malformations born to participants will be reported. Major congenital malformations are abnormalities of body structure or function that are present at birth and are of prenatal origin. Major congenital malformations include structural changes that have significant medical, social or cosmetic consequences for the affected individual, and typically require medical intervention (for example, cleft lip and spina bifida).
Percentage of Newborns Small for Gestational age (SGA) born to Participants | At birth
  Percentage of newborns small for gestational age (SGA) born to participants will be reported. Small for gestational age (SGA) means newborns that are smaller in size than normal for the gestational age (weight below the tenth percentile for the gestational age using Rwandan standards).
Percentage of Newborns with Low Birth Weight born to Participants | At birth
  Percentage of newborns with low birth weight born to participants will be reported. Low birth weight newborns are babies, weighing less than 2500 grams at birth (regardless of child's sex).
Percentage of Newborns with Preterm Birth born to Participants | At birth
  Percentage of newborns with preterm birth born to participants will be reported. Preterm birth means neonates born at less than 37 weeks' gestation.
Percentage of Neonatal Deaths in Neonates Born to Participants | Up to 28 days
  Percentage of neonatal deaths in neonates born to participants will be reported. Neonatal deaths mean neonate dying in the first 28 days of life.
Percentage of Infants (of Participants) who Fail to Thrive | From birth up to 14 weeks of age
  Percentage of infants (of participants) who fail to thrive will be reported. Failure to thrive means weight for age deceleration through at least 2 centile spaces on growth chart of infants or as defined according to Rwandan standards.

SECONDARY OUTCOMES:
Percentage of Participants (Pregnant Women) with Serious Adverse Events (SAEs) for Group A and B | Up to 6 weeks post-partum or post-pregnancy termination, whichever occurs earlier
  A SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Percentage of Participants (Pregnant Women) with SAEs for Subset of Group A and B | Up to 365 days or 1 year post dose
  A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above
Percentage of Newborns (Born to Participants) with SAEs | From birth up to 14 weeks of age
  A SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Percentage of Participants with Solicited Local and Systemic Adverse Events (AEs) | 7 Days after each vaccination (up to Day 64)
  Solicited local AEs: pain/tenderness, erythema, and induration/swelling. Solicited systemic AEs: headache, fatigue, myalgia, arthralgia, chills and fever.
Percentage of Participants with Unsolicited AEs | 28 Days after each vaccination (up to Day 85)
  Unsolicited AEs will include all AEs for which the participant is not specifically questioned in the participant diary.
Percentage of Participants with Normal Delivery | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with normal delivery will be reported.
Percentage of Participants with Caesarian Section | Up to 6 weeks post-completion/termination of pregnancy
  Percentage of participants with caesarian section will be reported.
Percentage of Participants with Anti-Ebola virus (EBOV) Glycoprotein (GP) Binding Antibodies | Day 1 (pre-dose 1), Day 78 (21 days post-dose 2), at delivery (Group A subset only), and 1 year post-dose 1 (Day 365)
  Blood samples will be collected for analysis of binding antibodies against EBOV GP using Filovirus Animal Non-Clinical Group (FANG) enzyme-linked immunosorbent assay (ELISA).
Percentage of Infants (Born to Participants) with Anti-Ebola virus (EBOV) Glycoprotein (GP) Binding Antibodies | From birth up to 14 weeks of age
  Blood samples will be collected from infants at 14 weeks of age for analysis of binding antibodies against EBOV GP using Filovirus Animal Non-Clinical Group (FANG) enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (3):
- Rwanda (3):
  - Gihundwe District Hospital, Cuangugu
  - Gisenyi Hospital, Gysenyi
  - Center for Family Health Research/Project San Francisco, Kigali

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Nyombayire J, Ingabire R, Mazzei A, Sharkey T, Umuhoza C, Mukamuyango J, Allen S, Tichacek A, Parker R, Wall KM, Katwere M, Keshinro B, Gaddah A, Wang Y, Forcheh CA, McLean C, Oriol-Mathieu V, Luhn K, Robinson C, Karita E. Heterologous two-dose Ebola vaccine regimen in pregnant women in Rwanda: a randomized controlled phase 3 trial. Nat Med. 2025 Nov;31(11):3899-3906. doi: 10.1038/s41591-025-03932-z. Epub 2025 Sep 8. PMID 40921806
- [Derived] Karita E, Nyombayire J, Ingabire R, Mazzei A, Sharkey T, Mukamuyango J, Allen S, Tichacek A, Parker R, Priddy F, Sayinzoga F, Nsanzimana S, Robinson C, Katwere M, Anumendem D, Leyssen M, Schaefer M, Wall KM. Safety, reactogenicity, and immunogenicity of a 2-dose Ebola vaccine regimen of Ad26.ZEBOV followed by MVA-BN-Filo in healthy adult pregnant women: study protocol for a phase 3 open-label randomized controlled trial. Trials. 2022 Jun 20;23(1):513. doi: 10.1186/s13063-022-06360-3. PMID 35725488